CLINICAL TRIAL: NCT04880122
Title: Comparison of Dried Blood Spots and Venous Blood for the Detection of SARS-CoV-2 2 Antibodies in a Population of Nursing Home Residents.
Brief Title: Dried Blood Spots for SARS-CoV-2 Serology (COVID-19).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BC-07665
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease
Keywords: serology; dried blood spot; elderly; nursing home residents; COVID-19; antibodies; immunoglobins; serosurveillance; vaccination; enzyme-linked immunosorbent assay (ELISA)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nursing home residents/staff members (Experimental): Matched venous blood/dried blood spots collection in a single arm.
  Interventions: Diagnostic Test: Dried blood spot and venous blood collection

INTERVENTIONS:
Diagnostic Test: Dried blood spot and venous blood collection — A paired venous blood and capillary blood sample (dried blood spot) were collected in every participant for validation purpose. Venous blood samples were analyzed using a chemiluminescent microparticle immunoassay ( the Architect i2000sr Plus system, Abbott), as a reference. Dried blood spots (EUROIMMUN, PerkinElmer Health Sciences Inc., Lübeck, Germany) or (Whatman™, GE Healthcare Sciences, Cardiff, UK) were analyzed by means of a SARS-CoV-2 IgG ELISA (EUROIMMUN, PerkinElmer Health Sciences Inc., Lübeck, Germany).

SUMMARY:
This study aims to validate dried blood spots (DBS) for SARS-CoV-2 (Severe Acute Respiratory Syndrome 2) antibody detection in elderly individuals.

DETAILED DESCRIPTION:
In the current SARS-CoV-2 pandemic, testing for SARS-CoV-2 specific antibodies is paramount to monitor immune responses in post-authorization vaccination and sero-epidemiology studies. However, large scale and iterative serological testing by venipuncture in older persons can be challenging. Capillary blood sampled using a finger prick and collected on protein saver cards, i.e., dried blood spots (DBS), has already proven to be a promising alternative. However, elderly persons have a reduced cutaneous microvasculature, which may affect DBS-based antibody testing. Therefore, we aimed to evaluate the performance of DBS for the detection of SARS-CoV-2 antibodies in nursing homes residents. We collected venous blood and paired Whatman and EUROIMMUN DBS from nursing home residents, and from staff as a reference population. Venous blood samples were analyzed for the presence of SARS-CoV-2 IgG antibodies using the Abbot chemiluminescent microparticle immunoassay (CMIA). DBS were analyzed by the EUROIMMUN enzyme-linked immuno sorbent assay (ELISA) for SARS-CoV-2 IgG antibodies.

ELIGIBILITY:
Inclusion Criteria:

* nursing home staff and residents

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of DBS for SARS-CoV-2 antibody detection | baseline (single timepoint)
  Sensitivity and specificity analysis
Optimization of the cut-off for seropositivity. | baseline (single timepoint)
  Optimization of the manufacturer recommended cut-off for seropositivity in DBS.

CONTACTS AND LOCATIONS:
Overall Officials: Piet Cools, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No